CLINICAL TRIAL: NCT02799589
Title: Remifentanil-dexmedetomidine Anesthesia as an Alternative Anesthetic for Elective Pediatric Surgery: a Pilot Study.
Brief Title: Remifentanil-dexmedetomidine Anesthesia With a Caudal for Elective Surgery. (Remi-dex)
Acronym: Remi-dex
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty in recruitment
Sponsor: Mofya Diallo (Other)
Responsible Party: Sponsor-Investigator, Mofya Diallo, Principal Investigator, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00006472
Record Dates: First submitted 2016-06-06; First posted 2016-06-15 (Estimated); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Remifentanil; Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remifentanil-dexmedetomidine and caudal (Experimental): Anesthesia will be induced with inhaled sevoflurane which will be discontinued once IV access is obtained and the airway is secured with an endotracheal tube. Patients will receive remifentanil loading dose of 1mcg/kg over 1 min followed by an infusion (0.05-0.5 mcg/kg/min) and dexmedetomidine load at 1mcg/kg over 10 mins followed by and infusion (0.2-0.7 mcg/kg/hr) A caudal block with 0.2% ropivacaine will be performed in all patients for intraoperative and postoperative pain control.
  Interventions: Drug: Remifentanil; Drug: Dexmedetomidine; Drug: Ropivacaine

INTERVENTIONS:
Drug: Remifentanil — 1mcg/kg over 1 min followed by an infusion (0.05-0.5 mcg/kg/min)
  Other Names: Ultiva
Drug: Dexmedetomidine — 1mcg/kg over 10 mins followed by and infusion (0.2-0.7 mcg/kg/hr)
  Other Names: Precedex
Drug: Ropivacaine — Caudal anesthesia block with Ropivicaine 0.2% 1ml/kg injected into the caudal space
  Other Names: Naropin

SUMMARY:
This study intends to show the efficacy of remifentanil-dexmedetomidine infusions in combination with a caudal block for patients ages 1 year to 3 years old receiving elective surgery to investigate alternatives to the currently used volatile anesthetics.

DETAILED DESCRIPTION:
In light of the concern for potential anesthetic neurotoxicity in infants and toddlers, it is prudent to start investigating alternative methods to decrease the amount of volatile anesthetic being utilized in this patient population. The US Food and Drug Administration has been asked to evaluate the data showing the neurotoxic effects of multiple anesthetic agents in animal models and humans. These studies have shown that N-methyl-D-aspartate (NMDA) receptor blockers such as ketamine,and gamma-Aminobutyric acid receptor (GABA) modulators like benzodiazepines, nitrous, propofol, barbiturates and isoflurane have been shown to cause brain cell apoptosis in animal models.

Regional anesthesia provides both intraoperative and postoperative analgesia may play a major role in effectively reducing the amount of general anesthetic used. Caudal anesthesia has been proven be both safe, effective and is applied widely in the pediatric population.

Dexmedetomidine is a selective alpha2-adrenergic agonist that acts in the brainstem by inhibiting norepinephrine release. Dexmedetomidine is commonly used off-label, including use for duration greater than 24 hours and any use in pediatrics. Dexmedetomidine has relatively few adverse events when compared to other sedative agents, with hypotension and bradycardia being most common.

Remifentanil has a rapid onset, rapid offset, small volume of distribution, rapid clearance, and a short elimination half-life, It may be a useful anesthetic for pediatric outpatient surgery.

While the current standard of care involves a volatile general anesthetic with a caudal block, anesthesiologists have alternative methods that can be utilized to allow an elective surgery to be performed. In summary, this study intends to show the efficacy and safety of a remifentanil-dexmedetomidine infusion and caudal block for patients ages 1 year-3 years old receiving elective circumcision, hydrocele repair, orchidopexy, mild hypospadias or inguinal hernia repair. This alternative anesthetic is already being studied in children under 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 - 3 years undergoing urologic surgery (circumcision, hydrocele repair, orchidopexy, mild hypospadias) or inguinal hernia repair
* American Society of Anesthesiologist Physical Status (ASA-PS) I or II
* Eligible for caudal block
* Parental/legal guardian consents for study '

Exclusion Criteria:

* Allergy to remifentanil, dexmedetomidine or ropivacaine
* Family history of malignant hyperthermia
* Parental/legal guardian refusal
* ASA-PS ≥ 3
* Symptoms of upper respiratory infection (URI) within the 2 weeks prior to surgery
* Known spinal deformity, presence of sacral dimple, or signs of infection at the site of the caudal block (e.g. diaper rash, skin redness or tenderness).

Ages: 1 Year to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Number of patients requiring intervention for light anesthesia | 90-120 mins (length of surgery)
  Identified by patient movement, change in mean arterial pressure >80 at surgical incision, need to change anesthetic plan

SECONDARY OUTCOMES:
Time to recovery after anesthesia | 10 mins; 1- 4 hours
  Time from end of surgery to: extubation; time to discharge from post-anesthesia care unit (PACU)
Number of patients requiring rescue analgesia in PACU | 30 mins to 4 hours after surgery
  Use of Fentanyl, Morphine, Ketorolac in recovery unit,
Number of patients with pain after surgery | 1 to 4 hours
  Pain is assessed after recovery on Face, Legs, Activity, Cry, Consolability (FLACC) scale 0 to 10. Average score will be noted.
Number of patients with respiratory event | Anesthesia start to discharge from PACU usually 2- 6 hours
  Bronchospasm, laryngospasm and pulse oximetry desaturation to less than 90%

CONTACTS AND LOCATIONS:
Overall Officials: Mofya Diallo, MD, Principal Investigator — Children's National Research Institute

IPD SHARING:
Plan to Share IPD: No